CLINICAL TRIAL: NCT02530749
Title: Frailty as a Predictor of Neurosurgical Outcomes in Brain Tumor Patients
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 14-0579
Record Dates: First submitted 2015-08-10; First posted 2015-08-21 (Estimated); Last update posted 2019-07-11 (Actual); Status verified 2019-07

CONDITIONS: Brain Tumors
Keywords: Surgery; Frailty
MeSH Terms: conditions — Brain Neoplasms; Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Frailty as an adjunct to preoperative assessment of neurosurgical patients has never been evaluated. This study aims to determine if frailty predicts neurosurgical complications in brain tumor patients and enhances current perioperative risk models.

DETAILED DESCRIPTION:
Preoperative risk assessment is important, but inexact, in older patients because physiologic reserves are difficult to measure. This also makes an important difference related to brain tumor patients, who may be burdened with systemic disease, alterations in cognition, or affected by other comorbidities. When assessing quality of life for brain tumor patients, having a better predictor of postsurgical outcome would be beneficial in appropriately counseling these patients. Frailty is thought to estimate physiologic reserves, and its use has been found to predict postoperative complications, length of stay, and discharge to a skilled or assisted-living facility in neurosurgical patients. Frailty as an adjunct to preoperative assessment of neurosurgical patients has never been evaluated. This study aims to determine if frailty predicts neurosurgical complications in brain tumor patients and enhances current perioperative risk models.

ELIGIBILITY:
Inclusion Criteria:

* Adult
* Ambulatory (able to walk)
* Scheduled for neurosurgical resection of brain tumor

Exclusion Criteria:

* Parkinson disease
* Previous stroke
* Taking: carbidopa/levodopa, donepezil hydrochloride, or antidepressants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study includes patients 18 years and older with a history of brain tumor scheduled for elective resection of tumor. Patients have to be ambulatory and be able to complete the examination and obtain a Hopkins Frailty Score.
Sampling Method: Non-Probability Sample
Enrollment: 265 (Actual)
Dates: Start 2014-04; Primary Completion 2018-12 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Number of patients with a Complication risk | 30 days
  Number of patients with a complication risk based on a Hopkins Frailty Score (HFS).

SECONDARY OUTCOMES:
Length of stay based on a Hopkins Frailty Score (HFS). | 30 days
  Number of patients with a prolonged length of stay based on a Hopkins Frailty Score (HFS).
Number of patients Discharge to a skilled or assisted-living facility | 30 days
  Number of patients discharged to a skilled or assisted-living facility based on a Hopkins Frailty Score (HFS).

CONTACTS AND LOCATIONS:
Overall Officials: D. R. Ormond, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States